CLINICAL TRIAL: NCT01830595
Title: Recombinant Lactoferrin to Reduce Immune Activation and Coagulation Among HIV Positive Patients
Brief Title: Lactoferrin Treatment in HIV Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jason Baker (Other)
Collaborators: Ventria Bioscience (Industry)
Responsible Party: Sponsor-Investigator, Jason Baker, Associate Professor of Medicine, Hennepin Healthcare Research Institute
Organization: Hennepin Healthcare Research Institute (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PCC-006
Record Dates: First submitted 2013-04-10; First posted 2013-04-12 (Estimated); Results first posted 2018-09-18 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recombinant Lactoferrin (Active Comparator): Recombinant lactoferrin will be administered by mouth twice daily
  Interventions: Drug: Recombinant Lactoferrin
- Placebo (Placebo Comparator): Matched placebo will be administered by mouth twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Recombinant Lactoferrin
  Arms: Recombinant Lactoferrin
Drug: Placebo
  Arms: Placebo

SUMMARY:
Our general goal is to evaluate the potential effectiveness of recombinant lactoferrin (1500mg bid) for reducing inflammation among HIV positive participants.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-positive participants receiving Antiretroviral Therapy (ART) for >1 year
2. HIV RNA level <200 copies/mL for at least 6 months (≥2 separate values)
3. Age >40 years

Exclusion Criteria:

1. Prior cardiovascular disease or stroke
2. Diabetes
3. Rheumatologic Diseases
4. Pregnancy
5. Chronic kidney disease, stage IV or V (creatinine clearance <30 mL/min/1.73m2)
6. Cirrhosis or end-stage liver disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason V Baker, MD, MS, Principal Investigator — Hennepin Healthcare Research Institute
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Sortino O, Hullsiek KH, Richards E, Rupert A, Schminke A, Tetekpor N, Quinones M, Prosser R, Schacker T, Sereti I, Baker JV. The Effects of Recombinant Human Lactoferrin on Immune Activation and the Intestinal Microbiome Among Persons Living with Human Immunodeficiency Virus and Receiving Antiretroviral Therapy. J Infect Dis. 2019 May 24;219(12):1963-1968. doi: 10.1093/infdis/jiz042. PMID 30721997

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant was administratively withdrawn prior to receiving medication.
Groups:
- Placebo First Then Lactoferrin: Participants receive placebo during first period, then Lactoferrin in second period after washout.
- Lactoferrin First Then Placebo: Participants receive Lactoferrin during first period, then placebo in second period after washout.
Period: First Period
Arm/Group | Placebo First Then Lactoferrin | Lactoferrin First Then Placebo
Started | 26 | 28
Received at Least One Dose | 26 | 28
Completed | 25 | 25
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3
Period: Washout
Arm/Group | Placebo First Then Lactoferrin | Lactoferrin First Then Placebo
Started | 25 | 25
Completed | 23 | 23
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 2 | 2
Period: Second Period
Arm/Group | Placebo First Then Lactoferrin | Lactoferrin First Then Placebo
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive placebo first and active drug first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.6 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 39
  Hispanic | 2
  African American | 11
  Other | 2
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm HG] — Population: All 54 participants started the first period, not all participants started the second period. Across both periods of treatment a total of 51 participants started Lactoferrin treatment and 49 participants started placebo treatment.
  mm HG
    At Enrollment | 79.5 (10.5)
    Beginning of Placebo Treatment: number analyzed (Participants) | 49
    Beginning of Placebo Treatment | 78.6 (9.9)
    Beginning of Lactoferrin: number analyzed (Participants) | 51
    Beginning of Lactoferrin | 79.3 (10.2)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] — Population: All 54 participants started the first period, not all participants started the second period. Across both periods of treatment a total of 51 participants started Lactoferrin treatment and 49 participants started placebo treatment.
  mm Hg
    At Enrollment | 129.7 (15.4)
    Beginning of Placebo Treatment: number analyzed (Participants) | 49
    Beginning of Placebo Treatment | 128.0 (14.9)
    Beginning of Lactoferrin Treatment: number analyzed (Participants) | 51
    Beginning of Lactoferrin Treatment | 127.8 (15.6)
Weight [Mean (Standard Deviation); unit: pounds] | 190.0 (38.1)
Interleukin-6 and D-Dimer Score [Mean (Standard Deviation); unit: scores on a scale] — The IL-6 & D-dimer score is defined as: 0. 33*log2 IL-6 + 0.16*log2 D-dimer, where IL-6 is measured in pg/mL and D-dimer in ug/mL. Since the biomarkers are on the log2 scale, associations of risk with the IL-6 & D-dimer score are interpreted as "Hazard Ratio (HR)(event) per doubling of IL-6 and D-dimer", or "HR(event) per 20% increase in IL-6 and D-dimer"; the score itself is unitless.
  Among the 3766 study participants for whom the score was developed, the min was -1.7, the max was 2.5.
  Higher scores are worse. Population: All 54 participants started the first period, not all participants started the second period. Across both periods of treatment a total of 51 participants started Lactoferrin treatment and 49 participants started placebo treatment.
  scores on a scale
    At Enrollment | -0.00 (0.38)
    Beginning of Placebo Treatment: number analyzed (Participants) | 49
    Beginning of Placebo Treatment | 0.02 (0.39)
    Beginning of Lactoferrin Treatment: number analyzed (Participants) | 51
    Beginning of Lactoferrin Treatment | -0.02 (0.45)
Small Artery Elasticity [Mean (Standard Deviation); unit: mL/mmHg x 100] — Population: All 54 participants started the first period, not all participants started the second period. Across both periods of treatment a total of 51 participants started Lactoferrin treatment and 49 participants started placebo treatment.
  mL/mmHg x 100
    At Enrollment | 6.49 (2.91)
    Beginning of Placebo Treatment: number analyzed (Participants) | 49
    Beginning of Placebo Treatment | 6.79 (3.04)
    Beginning of Lactoferrin Treatment: number analyzed (Participants) | 51
    Beginning of Lactoferrin Treatment | 6.61 (2.87)
Large Artery Elasticity [Mean (Standard Deviation); unit: mL/mmHg x 10] — Population: All 54 participants started the first period, not all participants started the second period. Across both periods of treatment a total of 51 participants started Lactoferrin treatment and 49 participants started placebo treatment.
  mL/mmHg x 10
    At Enrollment | 16.77 (5.74)
    Beginning of Placebo Treatment: number analyzed (Participants) | 49
    Beginning of Placebo Treatment | 17.02 (5.56)
    Beginning of Lactoferrin Treatment: number analyzed (Participants) | 51
    Beginning of Lactoferrin Treatment | 16.89 (5.48)
Monocyte CD16+ [Mean (Standard Deviation); unit: percent of total monocyte population] — Population: All 54 participants started the first period, not all participants started the second period. Across both periods of treatment a total of 51 participants started Lactoferrin treatment and 49 participants started placebo treatment.
  percent of total monocyte population
    At Enrollment | 10.55 (7.11)
    Beginning of Placebo Treatment: number analyzed (Participants) | 49
    Beginning of Placebo Treatment | 10.41 (7.56)
    Beginning of Lactoferrin Treatment: number analyzed (Participants) | 51
    Beginning of Lactoferrin Treatment | 11.96 (9.56)
sCD163 [Mean (Standard Deviation); unit: mg/L] — Population: All 54 participants started the first period, not all participants started the second period. Across both periods of treatment a total of 51 participants started Lactoferrin treatment and 49 participants started placebo treatment.
  mg/L
    At Enrollment | 0.21 (0.12)
    Beginning of Placebo Treatment: number analyzed (Participants) | 49
    Beginning of Placebo Treatment | 0.23 (0.15)
    Beginning of Lactoferrin Treatment: number analyzed (Participants) | 51
    Beginning of Lactoferrin Treatment | 0.19 (0.10)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Side Effect, Adverse Event, and Serious Adverse Event
Description: Self reported side effects and/or Division of AIDS (DAIDS) criteria will be used for grading adverse events (serious and non-serious)
Time Frame: During 3 months on Lactoferrin or Placebo (and following washout period)
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Matched placebo will be administered by mouth twice daily
  Placebo
- Recombinant Lactoferrin: Recombinant lactoferrin will be administered by mouth twice daily
  Recombinant Lactoferrin
Arm/Group | Placebo | Recombinant Lactoferrin
Number analyzed (Participants) | 54 | 54
Participants
  At least one side effect | 20 | 17
  At least one adverse event (includes SAE) | 12 | 11
  At least one Serious Adverse Event | 5 | 1

2. Primary Outcome: IL-6 & D-dimer Score Changes From Baseline to 3 Months (or Month 5 to Month 8)
Description: The IL-6 & D-dimer score is defined as: 0. 33*log2 IL-6 + 0.16*log2 D-dimer, where IL-6 is measured in pg/mL and D-dimer in ug/mL. Since the biomarkers are on the log2 scale, associations of risk with the IL-6 & D-dimer score are interpreted as "HR(event) per doubling of IL-6 and D-dimer", or "HR(event) per 20% increase in IL-6 and D-dimer"; the score itself is unitless.
  Among the 3766 study participants for whom the score was developed, the min was -1.7, the max was 2.5.
  Higher scores are worse.
Time Frame: 3 months (Baseline to Month 3 or Month 5 to Month 8)
Population: 45 participants contributed data during phase two. Participants had to attend the first visit (baseline or month 5) and also one follow-up visit in order to contribute data to the analyses.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Recombinant Lactoferrin
Number analyzed (Participants) | 45 | 45
score on a scale | -0.02 (0.39) | 0.06 (.36)
Statistical Analysis 1: Comparison: Placebo vs Recombinant Lactoferrin; Test type: Superiority; p = 0.38, t-test, 2 sided

3. Primary Outcome: Number of Participants Taking Medication as Assigned
Description: Number of participants taking medication as assigned at 3 months
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Recombinant Lactoferrin
Number analyzed (Participants) | 44 | 41
Participants | 40 | 38

4. Other Pre Specified Outcome: Activated Monocyte Phenotype (CD16+)
Description: The change in CD16+ monocyte subsets will be compared between active and placebo treatment phases. During both the active and placebo treatment phase, all relevant time points are used in calculation of change (i.e., baseline, month 1 and month 3 for phase 1; and similarly months 5, 6 and 8 for phase 2).
Time Frame: 3 months
Population: 45 participants contributed data during phase two. Participants had to attend the first visit (baseline or month 5) and also one follow-up visit in order to contribute data to the analyses. Fewer participants had pre-drug and post-drug cells collected so numbers are less than 45 for this measure.
Measure: Mean (Standard Deviation); unit: percent of total monocyte population
Arm/Group | Placebo | Recombinant Lactoferrin
Number analyzed (Participants) | 40 | 39
percent of total monocyte population | -0.45 (5.44) | -1.42 (9.26)
Statistical Analysis 1: Comparison: Placebo vs Recombinant Lactoferrin; Test type: Superiority; p = 0.55, t-test, 2 sided

5. Other Pre Specified Outcome: sCD163
Description: The change in blood levels of sCD163 will be compared between active and placebo treatment phases. During both the active and placebo treatment phase, all relevant time points are used in calculation of change (i.e., baseline, month 1 and month 3 for phase 1; and similarly months 5, 6 and 8 for phase 2).
Time Frame: 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Placebo | Recombinant Lactoferrin
Number analyzed (Participants) | 45 | 45
mg/L | -0.01 (0.06) | 0.03 (0.11)
Statistical Analysis 1: Comparison: Placebo vs Recombinant Lactoferrin; Test type: Superiority; p = 0.10, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | Placebo | Recombinant Lactoferrin
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/54
Serious Adverse Events (participants affected / at risk) | 5/54 | 1/54
Other Adverse Events (participants affected / at risk) | 10/54 | 10/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=54) | Recombinant Lactoferrin (N=54)
Hospitalization due to altered mental status (Psychiatric disorders) | 1 | 0
Hospitalization due to chest pain (Cardiac disorders) | 1 | 0
Hospitalization due to COPD (Respiratory, thoracic and mediastinal disorders) | 1 | 0
hospitalization for confusion, disorientation, shakiness, unsteady gait and vomiting (General disorders) | 1 | 0
Hospitalization for drug use (Nervous system disorders) | 1 | 0
Hospitalized for syncope episode (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=54) | Recombinant Lactoferrin (N=54)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Decreased appetite (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Insomnia (Nervous system disorders) | 1 | 0
Elevated CK (Musculoskeletal and connective tissue disorders) | 1 | 1
Elevated AST (General disorders) | 1 | 0
Skin infection (Infections and infestations) | 1 | 0
Bone (Musculoskeletal and connective tissue disorders) | 0 | 1 — broke left arm
Fatigue, cough and sore throat (Infections and infestations) | 0 | 1
Bone spur on spine (Musculoskeletal and connective tissue disorders) | 0 | 1
surgery on rotator cuff (Musculoskeletal and connective tissue disorders) | 0 | 1
torn rotator cuff (Musculoskeletal and connective tissue disorders) | 0 | 1
tinnitus (Ear and labyrinth disorders) | 0 | 1
right leg pain (Musculoskeletal and connective tissue disorders) | 0 | 1
nausea (General disorders) | 1 | 0
abdominal pain (General disorders) | 1 | 0
Cough and respiratory congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper Respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus Infection (Infections and infestations) | 1 | 0
Sinus pain and congestion (Infections and infestations) | 1 | 0
Cough, congestion, sinus pressure, fatigue (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-03-25): https://cdn.clinicaltrials.gov/large-docs/95/NCT01830595/Prot_SAP_ICF_000.pdf